CLINICAL TRIAL: NCT07169435
Title: Enhanced Reproductive Efficiency: Shorter Time to Pregnancy After Hysteroscopic-Assisted Novel Transvaginal Repair
Status: Completed | Type: Observational
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: (GKLW)2018-23
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Uterine Caesarean Scar Defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hysteroscopic-assisted novel transvaginal repair: Traditional transvaginal repair (TTR) procedure mainly involves two steps: the obvious scar-like defect excision and the full-thickness myometrial closure, which maybe form a new scar defect due to the uncertain scar healing process.
- Traditional transvaginal repair: Hysteroscopic-assisted novel transvaginal repair (NTR) surgery does not need to remove the original scar defect. Instead, suture was used to interruptedly suture the myometrium at the upper and lower margins of the scar to close the niche or reduce its size, which retains the integrity of the myometrium.

SUMMARY:
To investigate whether a novel hysteroscopic-assisted transvaginal repair technique results in a shorter time to pregnancy and superior fertility outcomes compared to traditional transvaginal repair.

ELIGIBILITY:
Inclusion Criteria:

Patients with a large niche (defined as niche with a depth of >50% of the myometrial thickness and a residual myometrial thickness (RMT) ≤3mm) Patients have fertility requirements Patients were aged between 18 and 48 years Patients who requested transvaginal surgery (the final decision about operation method was made by the patient (shared decision making))

Exclusion Criteria:

Patients with a narrow vaginal canal or any evidence of severe pelvic adhesion around the uterus Patients with post-operative biopsy-proven atypical endometrial hyperplasia and endometrial cancer

Ages: 18 Years to 48 Years | Sex: Female
Age Groups: Adult
Study Population: This prospective cohort study was conducted between May 2019 and May 2023 at Department of Gynecology and Obstetrics, International Peace Maternity and Child Health Hospital (IPMCH), Jiao Tong University School of Medicine, Shanghai, China.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
the median time to pregnancy following surgery | 2 years
  It is the time point at which half of the patients in the study who attempted to conceive after surgery had successfully become pregnant, and the other half had not

CONTACTS AND LOCATIONS:
Locations (1):
- International Peace Maternity and Child Health Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No